CLINICAL TRIAL: NCT02030925
Title: A Phase 2a Study to Evaluate the Effect of IW-3718 Administered Orally for 4 Weeks in Patients With GERD Not Completely Responsive to Proton Pump Inhibitors
Brief Title: Ph2a Study to Evaluate IW-3718 in Patients With Gastroesophageal Reflux Not Completely Responsive to Proton Pump Inhibitors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICP-3718-201
Record Dates: First submitted 2013-12-19; First posted 2014-01-09 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IW-3718 (Experimental): Twice a day
  Interventions: Drug: IW-3718
- Matching Placebo (Placebo Comparator): Twice a day
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: IW-3718
  Arms: IW-3718
Drug: Matching Placebo
  Arms: Matching Placebo

SUMMARY:
This study is meant to assess the effect of IW-3718 as an added treatment to ongoing once-daily protocol pump inhibitor (PPI) treatment for patients who continue to experience symptoms of their gastroesophageal reflux disease (GERD).

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 18 and 65 years of age at the Screening Visit; females must not be pregnant or must not be breastfeeding;
* Patient has a confirmed diagnosis of gastroesophageal reflux disease, must be currently taking a proton pump inhibitor (PPI), and must be experiencing GERD symptoms as specified by the protocol.

Exclusion Criteria:

* Patient may not meet any of the excluded conditions specified in the protocol;
* Patient is experiencing alarm symptoms such as GI bleeding, anemia, vomiting, dysphagia, or unexpected weight loss;
* Patient has a clinically significant hypersensitivity or allergies to any of the active ingredients or excipients in the study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Exploratory Endpoints - GERD Symptoms | Change from baseline: Treatment Period (weeks 1-4) compared with 2-week (baseline) Pretreatment Period

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Ironwood Investigational Site, North Little Rock, Arkansas
  - Ironwood Investigational Site, Anaheim, California
  - Ironwood Investigational Site, Monroe, Louisiana
  - Ironwood Investigational Site, Chesterfield, Michigan
  - Ironwood Investigational Site, Raleigh, North Carolina
  - Ironwood Investigational Site, Cleveland, Ohio
  - Ironwood Investigational Site, Chattanooga, Tennessee
  - Ironwood Investigational Site, Nashville, Tennessee
  - Ironwood Investigational Site, Logan, Utah
  - Ironwood Investigational Site, South Ogden, Utah